CLINICAL TRIAL: NCT03675451
Title: PSMA Imaging of Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1311014489
Record Dates: First submitted 2016-12-06; First posted 2018-09-18 (Actual); Results first posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: PET/CT; Imaging; Nuclear Medicine
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 89Zr-Df-IAB2M; gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Injection of study drug followed by PET/CT imaging.
  Optional but recommended 68Ga-PSMA-HBED-CC (5±2mCi) injection and PET/CT scan (1 to 3 hours after the injection) will also be performed prior to radical prostatectomy depending on subject's availability and compliance.
  Followed by prostatectomy
  Interventions: Drug: 89ZR-DF-IAB2M; Drug: 68Ga-PSMA-HBED-CC

INTERVENTIONS:
Drug: 89ZR-DF-IAB2M — injection of 10 milligrams of radioactive 89Zr-Df-IAB2M followed by PET/CT scan
Drug: 68Ga-PSMA-HBED-CC — Optional but recommended 68Ga-PSMA-HBED-CC (5±2mCi) injection and PET/CT scan (1 to 3 hours after the injection) will also be performed prior to radical prostatectomy depending on subject's availability and compliance.

SUMMARY:
The present study is a phase II, open label, single-center, non-randomized, single-dose study.

Twenty subjects in total will be enrolled at Weill Cornell Medical College (WCMC)/ NYPH.

The primary objective is to evaluate the ability of 89Zr-Df-IAB2M to detect localized, clinically significant (defined as: ≥ 0.5 cm3 with Gleason pattern ≥ 4) prostate cancer (PCa).

After the screening period (up to 28 days), each subject will be scheduled to receive 10 mg infusion of IAB2M conjugated with 2.5 mCi 89Zr-Df.

2 - 4 days post-infusion, subjects will undergo a 89Zr-Df-IAB2M PET/CT scan. Images read by a Nuc Med MD reporting: location, SUV and, if possible, size of all areas with abnormal uptake.

(they will also undergo a pelvic MRI if they have not obtained an MR image during the screening period or on day of infusion)

Optional but recommended 68Ga-PSMA-HBED-CC (5±2mCi) injection and PET/CT scan (1 to 3 hours after the injection) will also be performed prior to radical prostatectomy depending on subject's availability and compliance.

Patient will undergo radical prostatectomy after completion of above imaging procedures.

DETAILED DESCRIPTION:
The primary endpoint of this study is the proportion of subjects with PSMA-positive (identified by H&E staining and immunohistochemistry) "dominant" PC lesion(s) greater than 5mm in diameter, whose lesion(s) have been successfully identified by 89Zr-Df-IAB2M imaging. Because this is an exploratory pilot study, no formal sample size/power calculation is required. However, with a sample size of 20 patients in the study, a two-sided 95% confidence interval for the proportion of patients successfully imaged by 89Zr-Df-IAB2M can be constructed to be within ± 19.0% of the observed proportion of patients with successful imaging by 89Zr-Df-IAB2M. This calculation assumes an 89Zr-Df-IAB2M imaging-success proportion of 75%. All estimates from the study will serve as preliminary data (i.e., hypothesis-generating) for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed localized prostate cancer that are scheduled to undergo radical prostatectomy.
* Age >18 years.
* Patients must have laboratory values consistent with eligibility to undergo a radical prostatectomy:

  * creatinine less than or equal to 1.5 X upper limit of normal
  * creatinine clearance > 60 mL/min
* The effects of 89Zr-Df-IAB2M on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while her male partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Treatment or plans for treatment with radiation therapy, surgery, chemotherapy, or investigational therapy between the time of conventional imaging, 89Zr-Df-IAB2M PET/CT and the surgical resection used for the study evaluation.
* Transrectal prostate biopsy performed less than four weeks prior to 89Zr-Df-IAB2M administration.
* Uncontrolled illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas S Scherr, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Interventional: Injection of study drug followed by PET/CT imaging.
  Optional but recommended 68Ga-PSMA-HBED-CC (5±2mCi) injection and PET/CT scan (1 to 3 hours after the injection) will also be performed prior to radical prostatectomy depending on subject's availability and compliance.
  Followed by prostatectomy
  89ZR-DF-IAB2M: injection of 10 milligrams of radioactive 89Zr-Df-IAB2M followed by PET/CT scan
  68Ga-PSMA-HBED-CC: Optional but recommended 68Ga-PSMA-HBED-CC (5±2mCi) injection and PET/CT scan (1 to 3 hours after the injection) will also be performed prior to radical prostatectomy depending on subject's availability and compliance.
Period: Overall Study
Arm/Group | Interventional
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Interventional
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects With PSMA-positive (Prostate-specific Membrane Antigen) "Dominant" PC Lesion(s) Greater Than 5mm in Diameter, Whose Lesion(s) Have Been Successfully Identified by 89Zr-df-IAB2M PET/CT
Description: The number of subjects whose lesions have been successfully identified through 89Zr-df-IAB2M PET/CT will be ascertained using a combination of the descriptive statistics and lesion-based analysis, which both utilize multiple measurements
Time Frame: Up to 30 days pre-prostatectomy
Population: 19 of the 20 enrolled subjects were analyzed, as one of the 20 did not follow through with prostatectomy following 89Zr-df-IAB2M PET/CT, thus pathology is not available for 1 subject for this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- 89Zr-Df-IAB2M, mpMRI, Prostatectomy: 19 subjects were imaged with standard of care mpMRI injected with 10 milligrams of radioactive 89Zr-Df-IAB2M followed by PET/CT imaging, followed by prostatectomy
Arm/Group | 89Zr-Df-IAB2M, mpMRI, Prostatectomy
Number analyzed (Participants) | 19
Participants | 18
Statistical Analysis 1: Comparison: 89Zr-Df-IAB2M, mpMRI, Prostatectomy; Clopper-Pearson (Exact) 95% confidence interval to assess precision of finding; Test type: Other — Clopper-Pearson (Exact) 95% confidence interval to assess precision of finding; Proportion of Participants = 0.95, 95% CI 2-sided [0.74 to 0.99] — Clopper-Pearson (Exact) 95% confidence interval to assess precision of finding

2. Primary Outcome: The Number of Subjects With PSMA-positive "Dominant" PC Lesion(s) Greater Than 5mm in Diameter, Whose Lesion(s) Have Been Successfully Identified by 68Ga-PSMA-HBED-CC PET/CT
Description: The number of subjects with PSMA-positive (prostate-specific membrane antigen) "dominant" PC lesion(s) greater than 5mm in diameter, whose lesion(s) have been successfully identified by 68Ga-PSMA-HBED-CC PET/CT
Time Frame: Up to 30 days pre-prostatectomy
Population: 9 of the 20 enrolled subjects were analyzed, as only 9 subjects completed 68Ga-PSMA-HBED-CC PET/CT
Measure: Count of Participants; unit: Participants
Groups:
- 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy: A subset of 9 subjects were injected with 68Ga-PSMA-HBED-CC, followed by PET/CT scan (1 to 3 hours after the injection), performed prior to radical prostatectomy.
Arm/Group | 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy
Number analyzed (Participants) | 9
Participants | 9
Statistical Analysis 1: Comparison: 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy; Clopper-Pearson (Exact) 95% confidence interval to assess precision of finding; Test type: Other — Clopper-Pearson (Exact) 95% confidence interval to assess precision of finding; Proportion of Participants = 1.00, 95% CI 2-sided [0.66 to 1.00] — Clopper-Pearson (Exact) 95% confidence interval to assess precision of finding

3. Secondary Outcome: The Number of Clinically-significant Lesions Detected by 89Zr-df-IAb2M PET/CT
Time Frame: Up to 30 days pre-prostatectomy
Population: 19 of the 20 enrolled subjects were analyzed, as one of the 20 did not follow through with prostatectomy following study 89Zr-df-IAB2M PET/CT, thus pathology is not available.
Measure: Number; unit: Lesions
Arm/Group | 89Zr-Df-IAB2M, mpMRI, Prostatectomy
Number analyzed (Participants) | 19
Lesions | 22

4. Secondary Outcome: The Number of Clinically Significant Lesions Detected by 68Ga-PSMA-HBED-CC PET/CT
Description: Participants underwent 68Ga-PSMA-HBED-CC injection and PET/CT scan (1 to 3 hours after the injection),e performed prior to radical prostatectomy.
Time Frame: Up to 30 days pre-prostatectomy
Population: 9 of the 20 enrolled subjects were analyzed, as only 9 subjects completed 68Ga-PSMA-HBED-CC PET/CT
Measure: Number; unit: Lesions
Groups:
- 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy: A subset of 9 subjects were injected with 68Ga-PSMA-HBED-CC (5±2mCi), followed by PET/CT scan (1 to 3 hours after the injection), performed prior to radical prostatectomy.
Arm/Group | 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy
Number analyzed (Participants) | 9
Lesions | 10

5. Secondary Outcome: The Number of Clinically Significant Lesions Detected by mpMRI
Description: pre-prostatectomy standard of care mpMRI used to determine the number of clinically significant lesions
Time Frame: Up to 30 days pre-prostatectomy
Population: as for outcome 3
Measure: Number; unit: Lesions
Arm/Group | 89Zr-Df-IAB2M, mpMRI, Prostatectomy
Number analyzed (Participants) | 19
Lesions | 18

6. Secondary Outcome: The Number of Clinically Significant Lesions Detected by mpMRI in the Subset of Subjects Who Underwent 68Ga-PSMA-HBED-CC PET/CT
Description: The Number of Clinically Significant Lesions Detected by mpMRI in subjects who underwent 68Ga-PSMA-HBED-CC injection and PET/CT
Time Frame: Up to 30 days pre-prostatectomy
Population: 9 of the 20 enrolled subjects were analyzed, as only 9 subjects completed 68Ga-PSMA-HBED-CC PET/CT
Measure: Number; unit: Lesions
Arm/Group | 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy
Number analyzed (Participants) | 9
Lesions | 8

7. Secondary Outcome: The Number of Clinically Significant Lesions Detected by 89Zr-df-IAB2M PET/CT in the Subset of Subjects Who Underwent 68Ga-PSMA-HBED-CC PET/CT
Description: The Number of clinically significant lesions detected by 89Zr-df-IAB2M PET/CT in the subset of subjects who underwent 68Ga-PSMA-HBED-CC Injection and PET/CT
Time Frame: Up to 30 days pre-prostatectomy
Population: 9 of the 20 enrolled subjects were analyzed, as only 9 subjects completed 68Ga-PSMA-HBED-CC PET/CT
Measure: Number; unit: Lesions
Groups:
- 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy: A subset of 9 participants were injected with 68Ga-PSMA-HBED-CC (5±2mCi) followed by PET/CT imaging 1 to 3 hours after the injection. This preceded prostatectomy.
Arm/Group | 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy
Number analyzed (Participants) | 9
Lesions | 9

8. Secondary Outcome: The Number of Lesions Involved in Extra-prostatic Extension Identified Through in Vivo 89Zr-df-IAB2M PET/CT
Time Frame: Up to 30 days pre-prostatectomy
Population: 20 Subjects were injected with 10 milligrams of radioactive 89Zr-Df-IAB2M followed by PET/CT scan. 19 of those 20 completed prostatectomy and have pathology available for analysis.
Measure: Count of Units; unit: extra-prostatic lesions
Units Other Than Participants: extra-prostatic lesions
Arm/Group | 89Zr-Df-IAB2M, mpMRI, Prostatectomy
Number analyzed (Participants) | 19
Number analyzed (extra-prostatic lesions) | 12
extra-prostatic lesions | 9

9. Secondary Outcome: The Number of Lesions Involved in Extra-prostatic Extension Identified Through 68Ga-PSMA-HBED-CC PET/CT
Time Frame: Up to 30 days pre-prostatectomy
Population: A subset of 9 subjects were injected with 68Ga-PSMA-HBED-CC followed by PET/CT scan, prior to prostatectomy.
Measure: Count of Units; unit: extra-prostatic lesions
Units Other Than Participants: extra-prostatic lesions
Arm/Group | 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy
Number analyzed (Participants) | 9
Number analyzed (extra-prostatic lesions) | 4
extra-prostatic lesions | 4

10. Secondary Outcome: The Number of Occult Lymph Nodes Identified by in Vivo 89Zr-df-IAB2M PET/CT
Time Frame: Up to 30 days pre-prostatectomy
Population: as for outcome 3
Measure: Count of Units; unit: Occult Lymph Nodes
Units Other Than Participants: Occult Lymph Nodes
Groups:
- 89Zr-Df-IAB2M, mpMRI, Prostatectomy: 19 subjects were imaged with standard of care mpMRI injected with 10 milligrams of radioactive 89Zr-Df-IAB2M followed by PET/CT imaging, followed by prostatectomy
  A subset of 9 subjects were injected with 68Ga-PSMA-HBED-CC (5±2mCi), followed by PET/CT scan (1 to 3 hours after the injection), performed prior to radical prostatectomy.
Arm/Group | 89Zr-Df-IAB2M, mpMRI, Prostatectomy
Number analyzed (Participants) | 19
Number analyzed (Occult Lymph Nodes) | 10
Occult Lymph Nodes | 7

11. Secondary Outcome: The Number of Occult Lymph Nodes Identified by in Vivo 68Ga-PSMA-11 PET/CT
Time Frame: Up to 30 days pre-prostatectomy
Population: A subset of 9 of the 20 subjects were analyzed, as only 9 subjects completed 68Ga-PSMA-HBED-CC PET/CT. All 9 of those subjects had post-prostatectomy pathology for analysis.
Measure: Count of Units; unit: Occult Lymph Nodes
Units Other Than Participants: Occult Lymph Nodes
Groups:
- 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy: A subset of 9 participants were injected with 68Ga-PSMA-HBED-CC followed by PET/CT imaging 1 to 3 hours after the injection. This preceded prostatectomy.
Arm/Group | 89Zr-df-IAB2M, mpMRI, 68Ga-PSMA-11, and Prostatectomy
Number analyzed (Participants) | 9
Number analyzed (Occult Lymph Nodes) | 2
Occult Lymph Nodes | 2

12. Secondary Outcome: The Number of Observed or Reported Treatment-Emergent Adverse Events Following 89ZR-DF-IAB2M PET/CT (Positron Emission Tomography-Computed Tomography)
Description: All AEs, including unrelated AEs, expected, and unexpected AEs were included in the counts of adverse events
Time Frame: Up to 30 days pre-prostatectomy
Population: AEs were assessed for all 20 subjects who completed 89ZR-DF-IAB2M PET/CT.
Measure: Number; unit: Adverse Events
Groups:
- 89Zr-Df-IAB2M, mpMRI: 20 subjects were imaged with standard of care mpMRI injected with 10 milligrams of radioactive 89Zr-Df-IAB2M followed by PET/CT imaging.
  A subset of 19 subjects underwent prostatectomy following imaging
  A subset of 9 subjects were injected with 68Ga-PSMA-HBED-CC (5±2mCi), followed by PET/CT scan (1 to 3 hours after the injection), performed prior to radical prostatectomy.
Arm/Group | 89Zr-Df-IAB2M, mpMRI
Number analyzed (Participants) | 20
Adverse Events | 0

13. Secondary Outcome: The Number of Observed or Reported Treatment-Emergent Adverse Events Following 68Ga-PSMA-HBED-CC PET/CT
Description: All AEs, including unrelated AEs, expected, and unexpected AEs were included in the counts of adverse events
Time Frame: Up to 30 days pre-prostatectomy
Population: AEs were assessed for all 9 subjects who completed PET/CT.
Measure: Number; unit: Adverse Events
Arm/Group | 89Zr-Df-IAB2M, mpMRI
Number analyzed (Participants) | 9
Adverse Events | 0

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Groups:
- Interventional 89ZR-DF-IAB2M: 89ZR-DF-IAB2M: injection of 10 milligrams of radioactive 89Zr-Df-IAB2M followed by PET/CT scan
- 68Ga-PSMA-HBED-CC (5±2mCi): Injection of 68Ga-PSMA-HBED-CC (5±2mCi) injection and PET/CT scan (1 to 3 hours after the injection) will also be performed prior to radical prostatectomy depending on subject's availability and compliance.
Arm/Group | Interventional 89ZR-DF-IAB2M | 68Ga-PSMA-HBED-CC (5±2mCi)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/9
Other Adverse Events (participants affected / at risk) | 0/20 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/51/NCT03675451/Prot_SAP_000.pdf